CLINICAL TRIAL: NCT00259649
Title: Assessment and Prevention of Menstrual Migraine: Phase 1-prospective Survey of Self-identified Menstrual Migraine. Phase 2-prevention of Menstrual Migraine With Relpax
Brief Title: Prospective Survey of Menstrual Migraine & Prevention With Eletriptan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Dawn marcus, University of Pittsburgh
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 901423
Record Dates: First submitted 2005-11-26; First posted 2005-11-29 (Estimated); Results first posted 2011-07-04 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2011-06

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — eletriptan

INTERVENTIONS:
Drug: eletriptan — oral eletriptan 20 mg three times a day beginning 2 days before the expected onset of menstrual flow and continued for a total of 6 days
  Other Names: Relpax

SUMMARY:
Women are followed prospectively for 3 months, recording headaches, other symptoms, and menstrual periods. Those with menstrual migraine are treated perimenstrually with eletriptan for 3 months.

DETAILED DESCRIPTION:
Women are followed prospectively for 3 months, recording headaches, other symptoms, and menstrual periods. Those with menstrual migraine are treated perimenstrually with eletriptan for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* age 18-45 healthy menstruating female

Exclusion Criteria:

* cardiac or other conditions precluding use of eletriptan

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2004-08; Primary Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Marcus, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Eletriptan: Perimenstrual oral eletriptan 20 mg three times daily starting two days prior to the expected onset of menstruation and continued for a total of 6 days for 3 consecutive months
Period: Overall Study
Arm/Group | Eletriptan
Started | 71
Completed | 61
Not Completed | 10
Not completed — Lost to Follow-up | 7
Not completed — irregular menses | 3

BASELINE CHARACTERISTICS:
Arm/Group | Eletriptan
Number analyzed (Participants) | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 71
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 71

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Headache Index Score Among Patients
Description: Headache index is an average headache severity score recorded using a 0-10 severity scale recorded 4 times daily. Scores are averaged to produce an average severity score which can range between 0 (no headaches) to 10 (always a maximum severity headache). Change in headache activity was evaluated by comparing mean severity scores during the 3 months pre-intervention are compared with 3 months of preventive therapy
Time Frame: baseline to approximately three months
Measure: Mean (Standard Error); unit: headache index score
Arm/Group | Eletriptan
Number analyzed (Participants) | 71
headache index score | -1.52 (0.05)

ADVERSE EVENTS:
Description: 71 participants were enrolled in the study. Five did not receive treatment or attend their initial follow-up assessment. Therefore, AE data were only available for 66 participants.
Arm/Group | Eletriptan
Serious Adverse Events (participants affected / at risk) | 0/66
Other Adverse Events (participants affected / at risk) | 0/66

LIMITATIONS AND CAVEATS:
Relatively small sample size and open-label treatment limit Menstrual regulation by hormonal therapy might have affected treatment response;

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No